CLINICAL TRIAL: NCT02639780
Title: Biochemical Alterations of Stored Erythrocyte Membranes
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical Scientific Fund of the Mayor of Vienna (Other); European Society of Anaesthesiology (Other)
Responsible Party: Principal Investigator, David M Baron, MD, Assistant Professor, Medical University of Vienna
Other Study IDs: 1043/2015
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — packed red blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- healthy young female
  Interventions: Other: protein expression pattern of packed red blood cells
- healthy young male
  Interventions: Other: protein expression pattern of packed red blood cells
- healthy older female
  Interventions: Other: protein expression pattern of packed red blood cells
- healthy older male
  Interventions: Other: protein expression pattern of packed red blood cells
- obese older female
  Interventions: Other: protein expression pattern of packed red blood cells
- obese older male
  Interventions: Other: protein expression pattern of packed red blood cells

INTERVENTIONS:
Other: protein expression pattern of packed red blood cells — the proteome of packed red blood cells will be assessed at predefined time points

SUMMARY:
The investigators will define procoagulant properties of packed red blood cells and investigate whether packed red blood cells from certain donor populations are prone to induce procoagulant states.

ELIGIBILITY:
Inclusion Criteria:

* group 1: healthy female volunteers 18-35 y.o.
* group 2: healthy male volunteers 18-35 y.o.
* group 3: healthy female volunteers 36-60 y.o.
* group 4: healthy male volunteers 36-60 y.o.
* group 5: female volunteers 36-60 y.o., BMI 26-45
* group 6: male volunteers 36-60 y.o., BMI 26-45

Exclusion Criteria:

* age below 18 years
* age above 60 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: volunteers who will donate one unit of packed red blood cells
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
protein expression pattern | week 0
protein expression pattern | week 2
protein expression pattern | week 4
protein expression pattern | week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No